CLINICAL TRIAL: NCT00300989
Title: A Double-Blind,Randomised,Prospective Clinical Investigation to Compare Post-Operative Fracture Healing Using the Inion OTPS Biodegradable Fixation System Versus Conventional Metal Screws and Plates in the Treatment of Ankle Fractures.
Brief Title: Inion OTPS Biodegradable Fixation System for the Ankle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inion Oy (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D93-701 - 002
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Surgery

INTERVENTIONS:
Device: Inion OTPS Biodegradable Fixation System

SUMMARY:
The purpose of the investigation is to compare post-operative fracture and wound healing using Inion OTPS Biodegradable Fixation System implants versus Conventional metal implants.

ELIGIBILITY:
Inclusion Criteria:

* Distal fibular fracture including either instabile/dislocated Weber class B or any Weber class C fracture OR bimalloelar fracture with lateral malloelus fracture and medial malleolus fracture OR trimalleolar fracture with lateral and medial malleolus fractures and posterior malleolus fracture with less than 1/4 of the articulas surface fractured
* Fresh/acute fracture
* Aged between 18 and 60 years

Exclusion Criteria:

* Contraindication for the Inion OTPS Biodegradable Fixation System:Active or potential infection,patient's conditions, limited blood supply, insufficient quantity or quality of bone,where patient cooperation can not be quaranteed
* Multiple trauma
* Previous ankle fracture
* Pregnancy
* Bone malignancy
* Any clinically significant condition based on investigators judgement
* high-load bearing applications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2005-12; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Functional performance will be determined by using Kaikkonen Functional Scale (Kaikkonen et. al. 1994) and Olerud and Molander Ankle Score (Olerud and Molander 1984) at 12 months post-operatively.

SECONDARY OUTCOMES:
Sequential post-operative radiographs at 12 months post-operatively; Timepoints for returning to work and/or sport; Wound healing; SF-36 Questionnaire; Subjective pain evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ole Brink, Principal Investigator — Aarhus University Hospital; Terho Kainonen, Principal Investigator — Turku Universal Central Hospital; Geir Stray Andreassen, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Inion Oy, Tampere, Finland